CLINICAL TRIAL: NCT05586932
Title: The Effect of Iron Overload, Oxidative Stress and Dyslipidemia on Glucose Level and Thyroid Function in Patients With Abnormal Hemoglobinopathy
Brief Title: Oxidative Stress and Iron Overload in Patient With Abnormal Haemoglobinopathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Samar Gebril Mohamed Mahdy, Doctor, Assiut University
Other Study IDs: OxidativestressinabnormalHb
Record Dates: First submitted 2022-10-16; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Oxidative Stress in Patient With Haemoglobinopathy and Affect it of Endocrine System

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The effects of iron overload and oxidative stress and dyslipidemia on glucose level and thyroid function in patients with abnormal hemoglobinopathy. 2- Evaluation of MDA level as a marker of oxidative stress.

DETAILED DESCRIPTION:
Severe anemia due to defect in the synthesis of hemoglobin and hemolysis can endanger the life of β- thalassemia major (β-TM) patients and sickle cell anemia; therefore, the span and patient's quality of life is highly dependent on regular blood transfusion. Nonetheless, blood transfusion causes iron accumulation in the patients. Excess iron deposits in vital organs, such as liver, heart and endocrine glands, result in their malfunction. Endocrinopathies account as one of the most common iron overload complications. Oxidative stress is a major mechanism contributing to the progression of the disease in TDT. Iron overload enhances oxidative stress in patients with TDT. Iron is recognized to be a catalyst in developing reactive oxygen species (ROS).

MDA is an eosinophilic enol compound that reacts with the structural and functional cellular protein to generate toxic lipoxidation end product destined for cellular damage of the affected organs. It is used as a sensitive biomarker for oxidative stress. Disturbances in serum lipids and carbohydrates homoeostasis as well as OS were documented in β-TM and sickle cell anemia. Increase in serum levels total cholesterol (TC), low-density lipoprotein cholesterol (LDL-C) and decrease in high-density lipoprotein cholesterol (HDL-C) are the well-known causative factors and predictors of CHD development and endocrine abnormality

ELIGIBILITY:
Inclusion Criteria:

- age 18 and above.

-patients diagnosed according to physical examination and results of laboratory tests as beta thalassemia major. -patient under gradual blood transfusion and iron chelating therapy. -Gender and age matched healthy controls with normal serum lipid, glucose level and thyroid function will enrolled in this study as the control group

Exclusion Criteria:

* age under 18 years.
* patient diagnosed with DM or those taking pharmacological agents such as steroids, insulin and lipid lowering drugs

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will be done in Assiut University Hospital on 50 cases as Group (A): cases diagnosed as beta thalassemia major Group (B): healthy individuals (control)
  All patients will be subjected to full clinical history, examination and investigation. -investigation will include:
  * laboratory test:
  * CBC. -TSH, T4, T3. -serum oxidative stress marker (MDA).
  * glucose level.
  * cholesterol, triglycerides, HDl, LDL
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
correlation between oxidative stress and endocrine dysfunction in patients with hemoglubinopathy | 1 year
  1. The effects of iron overload and oxidative stress and dyslipidemia on glucose level and thyroid function in patients with abnormal hemoglobinopathy.

SECONDARY OUTCOMES:
Using of MDA level as a marker of oxidative stress | 1 year
  Malondialdehyde as a marker of oxidative stress

REFERENCES:
- See also: Endocrinopathies complicating transfusion-dependent hemoglobinopathy — https://pubmed.ncbi.nlm.nih.gov/32020146/
- See also: Pituitary Iron Deposition and Endocrine Complications in Patients with β-Thalassemia: From Childhood to Adulthood — https://pubmed.ncbi.nlm.nih.gov/32900239/
- See also: Sickle Cell Disease: Role of Oxidative Stress and Antioxidant Therapy — https://pubmed.ncbi.nlm.nih.gov/33669171/